CLINICAL TRIAL: NCT02276157
Title: A Prospective Randomized Trial of a New Multibending Versus Conventional Ultra-slim Endoscope for Direct Peroral Cholangioscopy Without Device Assistance
Brief Title: Direct Peroral Cholangioscopy by Using an Ultra-slim Upper Endoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Jong Ho Moon, Professor, Soonchunhyang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2014-07-026
Record Dates: First submitted 2014-10-21; First posted 2014-10-28 (Estimated); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Bile Duct Stricture; Choledocholithiasis
Keywords: cholangioscopy
MeSH Terms: conditions — Choledocholithiasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MB group (Experimental): Direct POC performed with third-generation prototype multibending ultra-slim endoscope (CHF-Y0010; Olympus Medical Systems, Co., Ltd., Tokyo, Japan)
  Interventions: Device: Direct peroral cholangioscopy
- Conventional group (Active Comparator): Direct POC performed with conventional ultra-slim endoscope (GIF-XP290N; Olympus Medical Systems, Co., Ltd., Tokyo, Japan)
  Interventions: Device: Direct peroral cholangioscopy

INTERVENTIONS:
Device: Direct peroral cholangioscopy — The multibending (MB) or conventional ultra-slim endoscope was inserted through the mouth. After facing the papillary orifice, the endoscope was inserted directly, without any accessories, into the distal bile duct. The second bending of the MB ultra-slim endoscope was kept in an upward angled position to achieve a more acute angle of the endoscope tip for entering the distal CBD. Then, the endoscope was pushed by steering the first bend into an upward angle ("α" shape) or the endoscope was pulled by steering the first bend into an upward angle and torqueing it counter-clockwise ("u" shape) for insertion into the distal CBD. If the distal bile duct was visualized on an endoscopic view, carbon dioxide insufflation was stopped. The endoscope was advanced into the hilum or the obstructed segment of the extrahepatic bile duct under fluoroscopic and endoscopic control. Then, the diagnostic and therapeutic interventions were performed during direct POC as necessary.

SUMMARY:
This study was aimed to to evaluate the efficacy of the new multibending ultra-slim endoscope compared with a conventional ultra-slim endoscope for free-hand insertion of an endoscope into the bile duct for direct POC.

DETAILED DESCRIPTION:
Currently available peroral cholangioscopy (POC) is a duodenoscopy-assisted procedure that does not involve directly inserting an endoscope into the biliary tree. A prototype multibending (MB) ultra-slim endoscope has been developed as a dedicated cholangioscope to overcome the technical difficulties of direct POC. In this study, the investigators evaluated the efficacy of the new MB ultra-slim endoscope compared with a conventional ultra-slim endoscope for free-hand insertion of an endoscope into the bile duct for direct POC without the assistance of accessories. The primary outcome was the technical success of free-hand insertion of the endoscope during direct POC, which was defined as successful insertion of the endoscope through the ampulla of Vater and advancement of the endoscope up to the bifurcation or to the obstructed segment of the biliary tree without any accessories within 15 min.

ELIGIBILITY:
Inclusion Criteria:

* biliary disease requiring diagnostic and/or therapeutic direct POC
* distal common bile duct (CBD) dilation > 8 mm
* previous sphincteroplasty, including major endoscopic sphincterotomy and/or endoscopic papillary balloon dilatation during a prior ERCP
* ability to provide informed consent

Exclusion Criteria:

* presence of any contraindication to ERCP
* bleeding tendency (international normalized ratio > 1.5 or platelet count < 50,000/ mm3)
* diffuse stricture of the distal CBD
* diagnosis of pancreatic cancer or tumor at the ampulla of Vater (AOV)
* altered gastrointestinal anatomy or significant duodenal obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2014-08; Primary Completion 2017-01 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
The technical success rate of free-hand insertion of an ultra-slim endoscope during direct POC | within 15 min after insertion of endoscope into the mouth
  successful insertion of the endoscope through the AOV and advancement up to the bifurcation or obstructed segment of the biliary tree, without any accessories

SECONDARY OUTCOMES:
Procedure time required for free-hand insertion | the time of oral intubation with the ultra-slim endoscope to the time of reaching the obstructed segment of the biliary tree or bifurcation, within 15 min after insertion of endoscope into the mouth
  Procedure time required for free-hand insertion
The technical success of diagnostic and therapeutic interventions | Within 24 hours after Completion of DPOC
  The technical success of diagnostic and therapeutic interventions
Adverse events related to direct POC | Within 7 days after DPOC
  perforation, cholangitis, pancreatitis, and air embolism

CONTACTS AND LOCATIONS:
Overall Officials: Jong Ho Moon, M.D., Ph.D., Principal Investigator — SoonChunHyang University School of Medicine
Locations (1):
- Soonchunhyang University Bucheon Hospital, Bucheon-si, South Korea

REFERENCES:
- [Background] Moon JH, Terheggen G, Choi HJ, Neuhaus H. Peroral cholangioscopy: diagnostic and therapeutic applications. Gastroenterology. 2013 Feb;144(2):276-282. doi: 10.1053/j.gastro.2012.10.045. Epub 2012 Nov 2. No abstract available. PMID 23127575
- [Result] Chen YK, Pleskow DK. SpyGlass single-operator peroral cholangiopancreatoscopy system for the diagnosis and therapy of bile-duct disorders: a clinical feasibility study (with video). Gastrointest Endosc. 2007 May;65(6):832-41. doi: 10.1016/j.gie.2007.01.025. PMID 17466202
- [Result] Choi HJ, Moon JH, Ko BM, Hong SJ, Koo HC, Cheon YK, Cho YD, Lee JS, Lee MS, Shim CS. Overtube-balloon-assisted direct peroral cholangioscopy by using an ultra-slim upper endoscope (with videos). Gastrointest Endosc. 2009 Apr;69(4):935-40. doi: 10.1016/j.gie.2008.08.043. PMID 19327480
- [Result] Moon JH, Ko BM, Choi HJ, Hong SJ, Cheon YK, Cho YD, Lee JS, Lee MS, Shim CS. Intraductal balloon-guided direct peroral cholangioscopy with an ultraslim upper endoscope (with videos). Gastrointest Endosc. 2009 Aug;70(2):297-302. doi: 10.1016/j.gie.2008.11.019. Epub 2009 Apr 25. PMID 19394010
- [Result] Moon JH, Ko BM, Choi HJ, Koo HC, Hong SJ, Cheon YK, Cho YD, Lee MS, Shim CS. Direct peroral cholangioscopy using an ultra-slim upper endoscope for the treatment of retained bile duct stones. Am J Gastroenterol. 2009 Nov;104(11):2729-33. doi: 10.1038/ajg.2009.435. Epub 2009 Jul 21. PMID 19623165
- [Result] Chen YK, Parsi MA, Binmoeller KF, Hawes RH, Pleskow DK, Slivka A, Haluszka O, Petersen BT, Sherman S, Deviere J, Meisner S, Stevens PD, Costamagna G, Ponchon T, Peetermans JA, Neuhaus H. Single-operator cholangioscopy in patients requiring evaluation of bile duct disease or therapy of biliary stones (with videos). Gastrointest Endosc. 2011 Oct;74(4):805-14. doi: 10.1016/j.gie.2011.04.016. Epub 2011 Jul 18. PMID 21762903